CLINICAL TRIAL: NCT03979300
Title: Learning Process of Fifth Years Medical Students During a Psychiatric Role Play : a Mixed Method Study
Brief Title: Learning Process of Fifth Years Medical Students During a Psychiatric Role Play
Status: Completed | Type: Observational
Sponsor: Institut Mutualiste Montsouris (Other)
Responsible Party: Sponsor
Other Study IDs: PSY-03-2018
Record Dates: First submitted 2018-08-03; First posted 2019-06-07 (Actual); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Educational
Keywords: Simulation training; Role-play; Psychiatry; Students; Medical; Psychology; Educational; Learning

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Other: Learning process during role play on psychiatric interview — Methodology: Mixed method study with:
  * Quantitative features:
    * Self-reported questionnaries : " Learning Effectiveness Inventory Scale " (18)
    * Sociodemographical data and others questions
  * Qualitative : Grounded Theory
    * Video-record of simulation and audio-record and briefing and debriefing, quoted with conversational analysis
    * Semi-structured interview of learners and teachers

SUMMARY:
This study aims to explore learning process in a role play for undergraduate students working on psychiatric interview. This study is one of the 3 studies included in a PhD on learning process during simulation training in psychiatry. The results of this 3 studies will aim at building a formative and summative assessment tool of competences specific to this pedagogic context

Methodology: Mixed method study with:

* Quantitative features:

  * Self-reported questionnaries : " Learning Effectiveness Inventory Scale "
  * Sociodemographical data and others questions
* Qualitative : Grounded Theory

  * Semi-structured interview of learners and teachers
  * Record of simulation and audio-record and briefing and debriefing (supplemented by quotation with conversational analysis (Rotterdam Interaction Analysis System, RIAS) for video)

DETAILED DESCRIPTION:
Since the end of the nineties, pedagogical transformations question traditional pedagogical system which favored a passive learning from master to student, trying to overcome classical " teaching paradigm" to " learning paradigm ". Despite several critics, the notion of " professional competence " emerges as one of the essential purpose of learning. Competence might be defined as " complex ability that professional built, starting from a specialized knowledge base, developed and controlled by a collegial peer who constitute the profession ", implying " a reflexive practice inside and after action " which creates or increases new competence in return.

However in french context, this paradigmatic revolution didn't really happened yet, including in psychiatry. Moreover, to our knowledge, there are no engineering didactic work on specific skills required by a physician (psychiatrist or not) should have in care of a patient with psychiatric disorders. For instance, skills required when a surgeon has to deliver a "clear, loyal and adjusted" information to a patient with a schizophrenia ; and try to get his or her agreement so as to operate a intestinal blockage? As a matter of facts, no integrated competence referential will be able to be a reference in this work.

In a report which is nowadays a reference for the faculties of medicine all over the world, the Royal College of Physicians and Surgeons of Canada (CRMCC) define a framework of essential skills that each physician have to control: medical expertise, erudition ; communicational and relational abilities; collaboration ; professionalism ; management; health promotion. In the French context, skills that each medical student have to provide for the psychiatric speciality are defined by 33 questions of national classifying exam (ECN). The " Psychiatry and Addictology Referential " points to medical students the reference knowledge to provide to respond to these questions during the challenge of ECN. But this referential doesn't explain skills, abilities and attitudes required with a patient with psychiatric disorders.

The places of providing essential skills defined by CRMCC applied in French psychiatry (as relational and communicational skills for instance) are thus often situated in others spaces. Realization of well supervised clerkship in psychiatry constitutes for example one of the privilege way of skills acquisition. Nonetheless in French context, all the undergraduate students can benefit from psychiatry during their clerkship; especially because of the rarefaction of well supervised internship (decreasing demography of psychiatrist), associated with increase number of medical student over the past few years. Moreover, realisation of an only internship can not include all the diversity of main family situation that should be known by each physician; mainly because of dichotomy of internship between adult and child and adolescent psychiatry, specific populations specific who go to different service according to there trouble (emergencies, closed unit, expert diagnosis centers…). Providing pedagogical tools allowing acquisition of basic skills, abilities and attitudes (complementary to knowledge and know-repeat) to care patient with psychiatric disorders seems thus interesting, for improving medical training.

Besides, assessment modalities determine for students work methodology and time involved in each learning, following Hawthorne effect. Assessments support learning assessed, involving long term memory, following " testing effect " ; and hierarchize planning of ulterior learning activities. Trials of ECN in this current shape will probably value acquisition of declarative knowledge for students who would like to succeed in the competition; to the detriment of know-how and life skills. These skills to care patients who suffer from psychiatric disorders won't be neither provided during a specialty residency, unless it might be especially oriented to psychiatry. Thus, it seems important to wider summative assessment modalities in psychiatry during undergraduate medical studies, so as to value acquisition of the wall skills required for a physician in care of a patient with psychiatric disorders. Which implies precise explanation of skills, abilities and attitudes needed, to balance success of ECN with their acquisition. In that context, simulation can offer a good response to this double aim : formative et summative. However, if some theorical approach are references to understand learning process in simulation, very few learning tool are validated in simulation, and none, to our knowledge, did a modelisation on learning process in psychiatric simulation for medical students.

ELIGIBILITY:
Inclusion Criteria:

FOR STUDENTS

* Age > to 18 years old
* Undergraduate medical fifth-years student of Paris Descartes University
* Studying on an integrated simulation training of Stomato, ORL, neurology and psychiatry
* Taking part in psychiatric simulation training associate with the course
* During university year 2017-2018
* French or English language

FOR TEACHERS

* Age > to 18 years old
* Teaching in psychiatric part to Undergraduate medical fifth-years student of Paris Descartes University in an integrated course of Stomato, ORL, neurology and psychiatry simulation training
* During university year 2017-2018
* French or English language

Exclusion Criteria:

* Refusal of agreement
* Undergraduate medical fifth-years student of Paris Descartes University, studying on an integrated course of stomatology, ORL, neurology and psychiatry, who didn't taking part in psychiatric simulation training associate with the course.
* Psychiatric teacher in Paris Descartes University who doesn't take part to psychiatric simulation training .

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Undergraduate medical fifth-years student of Paris Descartes University Teachers of Paris Descartes University
Sampling Method: Non-Probability Sample
Enrollment: 94 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2017-12-15 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Learning process | 6 weeks after learning process
  Learning process of 5th year medical students during simulation training in psychiatry.

SECONDARY OUTCOMES:
Factors influencing learning process | 6 weeks after learning process
  Factor influencing learning process of 5th year medical students during simulation training in psychiatry.
Satisfaction about learning | Immediately after simulation training
  Self-questionnaires : " Learning Effectiveness Inventory Scale "
Other questions (socio-demographic and specific to pedagogical design) | Immediately after simulation training
  Age, gender, previous simulation experience, and previous psychiatric experiences and psychiatric simulation experience, first, second and third specialty choice
RIAS video Cotations | 6 weeks after learning process
  Cotations of simulation video of students interviewed to face with their narratives
GT analysis of simulation video and audio-recorded briefing and debriefing | 6 weeks after learning process
  Cotations of simulation video and audio-recorded briefing and debriefing of students interviewed to face with their narratives

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Mutualiste Montsouris, Paris, Île-de-France Region, France